CLINICAL TRIAL: NCT02593058
Title: Positive Emotions Program for Schizophrenia (PEPS): A Randomized Controlled Study on Improving Pleasure and Motivation in Schizophrenia
Brief Title: Positive Emotions Program for Schizophrenia (PEPS)
Acronym: PEPS-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut et Haute Ecole de la Santé la Source (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Jérôme Favrod, Professor, Institut et Haute Ecole de la Santé la Source
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105319_163355 / 1
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Anhedonia; Apathy; Negative symptoms; Anticipatory pleasure; Savoring
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Anhedonia; Lethargy | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEPS+TAU (Experimental): Eight one-hour weekly sessions of Positive Emotions Program for Schizophrenia (PEPS) + Treatment as Usual (TAU)
  Interventions: Behavioral: Positive Emotions Program for Schizophrenia; Behavioral: Treatment As Usual
- Treatment As Usual (TAU) (Active Comparator): Treatment as usual - with no attempts to standardize this treatment as TAU is tailored to the patient's specific needs
  Interventions: Behavioral: Treatment As Usual

INTERVENTIONS:
Behavioral: Positive Emotions Program for Schizophrenia — Each session of PEPS includes relaxation-meditation exercise, review of homework task given during the previous session, exercises to challenge defeatist beliefs. According to the session's theme, participants learn skills to improve their anticipation or maintenance of pleasure such as savoring a pleasant experience, expressing emotions by increasing behavioral expression, capitalizing on positive moments, and anticipating pleasant moments. A simple homework task is assigned to be done between each session. The pedagogical concept underpinning the program was built according to Kolb and Kolb's model of experiential learning. The program uses a collaborative, egalitarian approach.
  Other Names: PEPS
  Arms: PEPS+TAU
Behavioral: Treatment As Usual — TAU consists of psychiatric management by a clinical team composed of at least one psychiatrist and a social worker and/or a psychiatric nurse with additional access to community treatment or hospital admission. Treatment involves antipsychotic medication, regular office-based or community contact with the clinical team for treatment monitoring, and socialization groups, therapy, and psychoeducational groups. No attempts have been made to standardize this treatment as TAU is tailored to the patient's specific needs.
  Other Names: TAU

SUMMARY:
This study evaluates the addition of a 8 session psychological program, called Positive Emotions Program for Schizophrenia (PEPS) to improve motivation and pleasure in adults with schizophrenia. Half of the participants will receive their usual treatment and PEPS in combination, while the other half will receive usual treatment only.

DETAILED DESCRIPTION:
Recent literature has distinguished the negative symptoms associated with a diminished capacity to experience (apathy, anhedonia) from those which are associated with a limited capacity for expression (emotional blunting, alogia). The apathy-anhedonia syndrome tends to be associated with a poorer prognosis than the symptoms related to diminished expression, suggesting that it is the more severe facet of the psychopathology. However the efficacy of drug-based treatments and psychological interventions on primary negative symptoms remains limited. There is a clear clinical need for developing treatments for negative symptoms.

The Positive Emotions Programs for Schizophrenia (PEPS) teaches skills to help overcome defeatist thinking and to increase the anticipation and maintenance of positive emotions. PEPS involves eight one-hour group sessions, administered using visual and audio materials as part of a PowerPoint presentation of slides projected onto a screen.

The goal of the study is to establish if PEPS is clinically effective by using a randomized, controlled and assessor-blind trial. A combination of PEPS plus treatment as usual will be compared to treatment as usual alone. Participants diagnosed with a schizophrenia spectrum disorder will undergo either intervention for eight weeks. Testing will evaluate individuals' current psychopathology and ability to savor pleasure and will be performed at the time of inclusion, at the end of the eight-week intervention and at six month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* a psychotic disorder according to ICD 10 (F20 or F25), diagnoses having been established by experienced clinicians;
* presenting a score of at least 2 on the overall SANS anhedonia scale;
* French-speaking;
* Ability to consent measured with the San Diego Brief Assessment of Capacity to Consent (UBACC)-a decisional capacity instrument.

Exclusion Criteria:

* evidence of organic brain disease, clinically significant concurrent medical ill/ness, or learning disability;
* no understanding of the study protocol as assessed with the San Diego Brief Assessment of Capacity to Consent (UBACC)-a decisional capacity instrument

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change on the composite score of apathy/avolition and anhedonia/asociality ot the Scale for the Assessment of Negative Symptoms (SANS). | Change from Baseline composite score at 2 months
  The Scale for the Assessment of Negative Symptoms (SANS) measures schizophrenia's deficit symptoms within the framework of schizophrenic disorders. It comprises 25 items, scored from 0 to 5. A definition of each item, including examples, facilitates a better understanding of the scale's content. The rating system is ordinal, from 0 (absent) to 5 (severe). The twenty-five items are grouped into five components: 1) withdrawal or emotional poverty; 2) alogia (lack of speech); 3) avolition and apathy (lack of energy, lack of initiative); 4) anhedonia and social withdrawal (loss of interests); 5) attention. The scale was translated into French with acceptable validity. The composite score for the avolition-apathy and anhedonia-social withdrawal scale will be used as the main outcome variable.

SECONDARY OUTCOMES:
Change on the Calgary Depression Scale for Schizophrenia (CDSS) | Change from Baseline CDSS score at 2 months
  The Calgary Depression Scale for Schizophrenia (CDSS) includes nine items: depression, hopelessness, self-depreciation, guilty ideas of reference, pathological guilt, morning depression, early wakening, suicide, and observed depression. This scale has been validated in French.
Change on the Savoring Belief Inventory (SBI) | Change from Baseline SBI total score at 2 months
  The Savoring Belief Inventory (SBI) is a self-reported scale for measuring beliefs about one's capacity for savoring things. The scale has twenty four items, including a positive scale (twelve items) and a negative scale (twelve items). The scale has good validity and a high test-re-test reliability. It measures a person's thinking regarding his/her capacity to savor positive experiences, in terms of past experiences, current experiences, and future anticipation. The total SBI score will be used as a secondary outcome variable.
Change on the Temporal Experience of Pleasure Scale (TEPS) | Change from Baseline TEPS scales at 2 months
  The Temporal Experience of Pleasure Scale (TEPS) is a self-reported scale and contains eighteen items included in two sub-scales: anticipatory pleasure (ten items) and consummatory pleasure (eight items). Items targeting anticipatory pleasure reflect the pleasure felt when anticipating a positive or pleasant stimulus. Items measuring consummatory pleasure refer to the direct pleasure experienced upon exposure to a stimulus. Items can be general or specific. The response to items falls on a six-point Likert scale from 1 (very false for me) to 6 (very true for me). This scale has been validated in French.
Change on the Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) | Change from Baseline ACIPS scales at 2 months
  The Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS) is designed to assess one's ability to experience pleasure in the interpersonal domain. It is a seventeen-item self-reported measure that consists of seven anticipatory and ten consummatory items. The ACIPS is scored on a six-point Likert scale, ranging from 1 (very false for me) to 6 (very true for me). The format is therefore quite similar to that of TEPS. The difference between the two scales lies mainly in terms of the items' content.
Change on the Social Functioning Scale (SFS) | Change from Baseline SFS at 8 months
  The Social Functioning Scale (SFS) is constructed to assess those areas of functioning that are crucial to the community maintenance of individuals with schizophrenia. This is a reliable, valid, sensitive instrument and responsive to change. This last scale will be completed by the case-manager of the participant.
Change on the Calgary Depression Scale for Schizophrenia (CDSS) | Change from Baseline CDSS score at 8 months
  The Calgary Depression Scale for Schizophrenia (CDSS) includes nine items: depression, hopelessness, self-depreciation, guilty ideas of reference, pathological guilt, morning depression, early wakening, suicide, and observed depression. This scale has been validated in French.
Change on the composite score of apathy/avolition and anhedonia/asociality ot the Scale for the Assessment of Negative Symptoms (SANS) | Change from Baseline composite score at 8 months
  The Scale for the Assessment of Negative Symptoms (SANS) measures schizophrenia's deficit symptoms within the framework of schizophrenic disorders. It comprises 25 items, scored from 0 to 5. A definition of each item, including examples, facilitates a better understanding of the scale's content. The rating system is ordinal, from 0 (absent) to 5 (severe). The twenty-five items are grouped into five components: 1) withdrawal or emotional poverty; 2) alogia (lack of speech); 3) avolition and apathy (lack of energy, lack of initiative); 4) anhedonia and social withdrawal (loss of interests); 5) attention. The scale was translated into French with acceptable validity. The composite score for the avolition-apathy and anhedonia-social withdrawal scale will be used as the main outcome variables.

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Favrod, Principal Investigator — Institut et Haute Ecole de la Santé la Source & Service de psychiatrie communautaire du Département de psychiatrie du Centre Hospitalier Universitaire Vaudois
Locations (1):
- Institut et Haute Ecole de la Santé la Source & Service de psychiatrie communautaire du Département de psychiatrie du Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Favrod J, Nguyen A, Fankhauser C, Ismailaj A, Hasler JD, Ringuet A, Rexhaj S, Bonsack C. Positive Emotions Program for Schizophrenia (PEPS): a pilot intervention to reduce anhedonia and apathy. BMC Psychiatry. 2015 Sep 29;15:231. doi: 10.1186/s12888-015-0610-y. PMID 26419356
- [Background] Favrod J, Giuliani F, Ernst F, Bonsack C. Anticipatory pleasure skills training: a new intervention to reduce anhedonia in schizophrenia. Perspect Psychiatr Care. 2010 Jul;46(3):171-81. doi: 10.1111/j.1744-6163.2010.00255.x. PMID 20591125
- [Background] Golay P, Thonon B, Nguyen A, Fankhauser C, Favrod J. Confirmatory Factor Analysis of the French Version of the Savoring Beliefs Inventory. Front Psychol. 2018 Feb 19;9:181. doi: 10.3389/fpsyg.2018.00181. eCollection 2018. PMID 29515496
- [Background] Chaix J, Golay P, Fankhauser C, Nguyen A, Gooding DC, Favrod J. Confirmatory Factor Analysis of the French Version of the Anticipatory and Consummatory Interpersonal Pleasure Scale. Front Psychol. 2017 Jul 28;8:1296. doi: 10.3389/fpsyg.2017.01296. eCollection 2017. PMID 28804473
- [Background] Nguyen A, Frobert L, McCluskey I, Golay P, Bonsack C, Favrod J. Development of the Positive Emotions Program for Schizophrenia: An Intervention to Improve Pleasure and Motivation in Schizophrenia. Front Psychiatry. 2016 Feb 17;7:13. doi: 10.3389/fpsyt.2016.00013. eCollection 2016. PMID 26924992
- [Result] Favrod J, Nguyen A, Chaix J, Pellet J, Frobert L, Fankhauser C, Ismailaj A, Brana A, Tamic G, Suter C, Rexhaj S, Golay P, Bonsack C. Improving Pleasure and Motivation in Schizophrenia: A Randomized Controlled Clinical Trial. Psychother Psychosom. 2019;88(2):84-95. doi: 10.1159/000496479. Epub 2019 Feb 18. PMID 30783071
- See also: Intervention description and materials — http://www.seretablir.net/outils-interventions/peps/